CLINICAL TRIAL: NCT06828575
Title: Evaluation of the Success of Artificial Intelligence Models in Interpreting Arterial Waveform Analysis Data
Status: Recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: mostcare
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Drug Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: predictions — predictions of learning language models

SUMMARY:
The goal of this observational study is to evaluate the ability of artificial intelligence (AI) models to interpret arterial waveform analysis data obtained from a hemodynamic monitoring system in adult patients undergoing elective surgery. The main questions it aims to answer are:

Can AI models (ChatGPT-4 and Gemini 2.0) accurately detect hemodynamic abnormalities in arterial waveform data? How well do AI-generated diagnoses align with expert anesthesiologist assessments? Are AI-generated treatment recommendations clinically appropriate?

Participants will:

Undergo standard hemodynamic monitoring with an arterial waveform analysis device (MostCare).

Have their anonymized hemodynamic data analyzed by AI models for abnormality detection, diagnosis suggestions, and treatment recommendations.

Have AI-generated results reviewed and validated by experienced anesthesiologists.

This study aims to assess whether AI models can serve as decision-support tools in perioperative and critical care settings by improving the interpretation of complex hemodynamic data, potentially enhancing patient safety, diagnostic accuracy, and clinical efficiency.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the ability of artificial intelligence (AI) models to interpret arterial waveform analysis data obtained from a hemodynamic monitoring system. The study will focus on assessing the accuracy of ChatGPT-4 and Gemini 2.0 in detecting hemodynamic abnormalities, providing diagnostic suggestions, and offering treatment recommendations based on arterial waveform data collected from elective surgical patients.

Background and Rationale Arterial waveform analysis is a critical component of advanced hemodynamic monitoring, providing real-time insights into cardiac output, vascular resistance, and volume status. These parameters are essential for guiding perioperative fluid management and optimizing hemodynamic stability in surgical and critically ill patients. While automated monitoring systems generate large amounts of data, the interpretation of these waveforms remains dependent on clinician expertise. The integration of AI-based decision-support tools in this context could enhance real-time clinical decision-making and reduce workload for healthcare providers.

Study Objectives

The primary objective of this study is to determine the ability of AI models to analyze arterial waveform data and detect clinically significant hemodynamic abnormalities. The secondary objectives are:

To assess the concordance between AI-generated diagnoses and expert anesthesiologist assessments.

To evaluate the clinical appropriateness of AI-generated treatment recommendations.

To explore the potential role of AI in clinical decision support systems for hemodynamic monitoring.

Study Design and Methodology

This study will be conducted at two tertiary-level healthcare institutions:

Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital Başakşehir Çam and Sakura City Hospital The study will include adult patients undergoing elective surgery who require intraoperative arterial waveform monitoring as part of routine perioperative care.

Data Collection Process Hemodynamic data will be collected from participants using the MostCare hemodynamic monitoring system, which is routinely used in perioperative settings.

Data collection will take place at three time points:

Pre-anesthesia (baseline hemodynamic status before induction) Post-anesthesia induction (after intubation, before surgical incision) Intraoperative period (during key surgical events requiring hemodynamic intervention) If an intervention needs according to arterial wave analysis we will also take data before and after intervention.

AI-Based Analysis

The collected arterial waveform data will be anonymized and processed by AI models (ChatGPT-4 and Gemini 2.0) to provide:

Abnormality detection - Identifying any deviations from normal hemodynamic parameters.

Diagnostic suggestions - Providing likely clinical diagnoses based on the waveform patterns.

Treatment recommendations - Suggesting possible interventions to optimize hemodynamic status.

Expert Validation AI-generated results will be independently reviewed by experienced anesthesiologists to assess their accuracy and clinical relevance.

The concordance between AI outputs and expert assessments will be statistically analyzed.

Outcome Measures

Primary Outcome:

Accuracy of AI models in detecting hemodynamic abnormalities compared to expert assessments.

Secondary Outcomes:

Concordance between AI-generated diagnoses and anesthesiologist diagnoses. Clinical appropriateness of AI-generated treatment recommendations compared to standard clinical practice.

AI models' potential role in enhancing clinical decision-making in perioperative hemodynamic management.

Ethical Considerations The study does not involve any additional interventions beyond routine clinical monitoring.

No patient-identifiable data will be used in AI model analysis. Informed consent will be obtained from all participants before enrollment. The study has been approved by the relevant ethics committees at both participating institutions.

Study Timeline Planned study duration: 6 months Estimated start date: February 15, 2025 Estimated completion date: August 15, 2025 Potential Impact

This study will provide valuable insights into the role of AI in automated hemodynamic monitoring and perioperative decision support. If successful, AI-driven analysis of arterial waveform data could:

Enhance patient safety through early detection of hemodynamic abnormalities. Improve efficiency by assisting anesthesiologists in data interpretation. Reduce workload for perioperative and critical care teams. Support future AI-based clinical decision-support tools for hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing elective surgery with arterial waveform monitoring as part of standard perioperative care
* Hemodynamic data successfully recorded using the MostCare hemodynamic monitoring system
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* Incomplete or corrupted hemodynamic data (e.g., signal artifacts preventing reliable analysis)
* Emergency surgery cases
* Patients with severe arrhythmias or hemodynamic instability that might interfere with arterial waveform interpretation
* Refusal to participate or withdrawal of consent
* Patients with contraindications to arterial catheterization (e.g., coagulopathy, severe peripheral vascular disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients (≥18 years old) undergoing elective surgery requiring intraoperative arterial waveform monitoring as part of routine perioperative care. The population will consist of patients from two tertiary-level hospitals where advanced hemodynamic monitoring with the MostCare system is regularly utilized.
  Participants will be selected based on their eligibility for continuous arterial pressure monitoring, ensuring a standardized dataset for AI analysis. The study population will represent a diverse range of surgical procedures, including but not limited to:
  General surgery (e.g., abdominal, hepatobiliary, colorectal procedures)
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 1 day
  Accuracy of AI models in detecting hemodynamic abnormalities (True or False).

SECONDARY OUTCOMES:
Concordance Between AI-Generated Diagnoses and Expert Anesthesiologist Diagnoses | 1 DAY
  AI-generated diagnostic suggestions will be compared with the final diagnosis made by anesthesiologists (True or False).
Clinical Appropriateness of AI-Generated Treatment Recommendations | 1 DAY
  The relevance and accuracy of AI-suggested treatments will be evaluated against standard clinical management (True or False).

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided